CLINICAL TRIAL: NCT02938104
Title: Multimodal Prehabilitation to Enhance Functional Recovery After Lung Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Franco Carli (Other)
Collaborators: Immunotec Inc. (Industry)
Responsible Party: Sponsor-Investigator, Franco Carli, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 14-193-GEN
Record Dates: First submitted 2016-02-02; First posted 2016-10-19 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prehabilitation (Experimental): Immediately after randomization, until surgery and to be continued for 8 weeks after surgery, patients in this arm will:
  1. Receive a personalized physical exercise program
  2. Receive nutritional counselling with whey protein isolate powder
  3. Receive relaxation techniques
  Interventions: Dietary Supplement: Whey Protein Isolate Powder; Behavioral: Physical Exercise Program; Behavioral: Relaxation Techniques
- Rehabilitation (Active Comparator): Patients in this arm will receive the same personalized physical exercise program, nutritional intervention and relaxation techniques as patient in the other arm but to be started after surgery.
  Interventions: Dietary Supplement: Whey Protein Isolate Powder; Behavioral: Physical Exercise Program; Behavioral: Relaxation Techniques

INTERVENTIONS:
Dietary Supplement: Whey Protein Isolate Powder — Nutritional counselling is given to patients to ensure their daily proteins and energy requirements are met. Whey Protein Isolate Posder (Immunocal) is provided.
  Immunocal (1.5g/kg PO (by mouth) per day in daily doses
Behavioral: Physical Exercise Program — Physical exercises personalized by a kinesiologist consisting of walking or stationary bike and elastic band exercises.
Behavioral: Relaxation Techniques — Relaxation techniques consisting of breathing exercises and using a relaxation CD

SUMMARY:
The investigators propose a randomized controlled study in patients undergoing lung resection for cancer to compare the impact of multimodal intervention composed of exercise, nutritional supplement and psychological well-being on functional exercise capacity. One group (rehabilitation group) will receive the multimodal intervention after surgery for 8 weeks; the other will start 4 weeks before surgery and continue for 8 weeks postop (prehabilitation group). In this case, both groups will be exposed to the program, which will be available to both groups postoperatively. One of the two groups will start this program 4 weeks before surgery and continue for 8 weeks postoperatively, and the other will start once they leave the hospital and continue for 8 weeks postoperatively.

DETAILED DESCRIPTION:
Interventions

The multidisciplinary program is composed of 3 elements: exercise, nutritional supplements and psychological coping strategies

Exercise program

Patients will be seen by a kinesiologist for a period of 1 hour and he/she will assess patients' mobility and capacity to undertake exercise, will prepare a personalized program and will explain and monitor the exercise program. Patients will be instructed on how to conduct aerobic exercise in the lab and at home, by either walking or cycling initially at 50% of the calculated heart rate reserve for 20 min three times per week, and this will be increased in stepwise increments by 10% each week, if tolerable.

Muscular resistance training will be also carried out 3 times a week to avoid muscle soreness. Persons will be instructed to do push-up, sit-ups, and standing strides (lunges) until volitional fatigue increasing this number to reach 12 repetitions. The resistance chosen for strengthening of biceps, deltoids and quadriceps will be based on what the person can lift to reach volitional fatigue with 8 repetitions.

Psychological program

It is expected that patients undergoing surgery for cancer are anxious with some component of depression. Since both anxiety and depression can influence the motivation to carry out social and functional activities, psychological strategies can be put in place to help patients to cope with the stress of surgery and disease. For this reason patients will be seen by a trained psychologist. Patients will receive a total of 1.5 hours of psychological intervention in the first session and more sessions if necessary.

In the first preoperative session, the first hour will address the patient's anxieties, coping strategies, and post-operative expectations, with the goal of optimizing psychological well-being & ways of coping with surgery. The importance of the patient's active participation in the healing process will also be discussed. The last thirty minutes will be devoted to teaching relaxation techniques and breathing exercises. Patients will be given a relaxation CD to take home for practice.

Nutritional supplementation

The nutritional status of patients affected by lung cancer is directly influenced by the presence of cancer, which impacts on all aspects of intermediary (protein, carbohydrate, lipid, trace element, vitamin) metabolism, and by other factors such as age, adjuvant cancer therapy and stage of the disease. The greater sensitivity of protein catabolism to nutritional support, in particular to amino acids, could have important implications for the nutritional management of these patients during the period of catabolic stress, with particular emphasis on substrate utilization and energy requirement.

The patients' nutritional status and dietary intake will be assessed by the nutritionist. Percentage of lean body mass and fat percentage will be measured. All patients will receive a daily dietary supplement known as whey protein (Immunocal, Immunotec ©). Special precautions will be considered if patients have specific medical conditions (e.g. diabetes).

ELIGIBILITY:
Inclusion Criteria:

* aged 18 and above
* referred electively for resection of malignant, non-metastasized lung lesion

Exclusion Criteria:

* persons with American Society of Anesthesiologists (ASA) health status class 4-5
* persons with co-morbid medical, physical, and mental abnormalities (e.g. dementia, disabling orthopedic and neuromuscular disease, psychosis), cardiac abnormalities, severe end-organ disease such as cardia failure, COPD, renal failure, sepsis, morbid obesity, anemia, and other conditions interfering with the ability to perform exercise at home or to complete testing procedures
* poor English or French comprehension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-08; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Six-minute walk test | 8 weeks after surgery
  The 6MWT evaluates the ability of an individual to maintain a moderate level of physical activity over a time period reflective of the activities of daily living. Subjects are instructed to walk back and forth, in a 20 m stretch of hallway, for six minutes, at a pace that would make them tired by the end of the walk; encouragement and feedback are given according to published guidelines.

SECONDARY OUTCOMES:
Health-related quality of life | 8 weeks after surgery
  The SF-36 incorporates behavioural functioning, subjective well-being and perceptions of health by assessing, on a 0 to 100 scale, eight health concepts: (1) Physical function (PF) -limitations in physical activities due to health problems; (2) Role physical (RP)-limitations in role activities due to physical health problems; (3) Role emotional (RE) -limitations in usual role activities due to emotional problems; (4) Social functioning (SF) -limitations in social activities due to health problems; (5) Bodily pain (BP)-pain; (6) General health (GH) -general health perceptions; (7) Vitality (VT) -energy and fatigue; and (8) Mental health (MH) -general mental health.
Quality of Life | 8 weeks after surgery
  The FACT-L (functional assessment of cancer therapy lung) and EQ-5D, both validated measures, will be used to assess quality of life.
Physical activity level | 8 weeks after surgery
  Physical activity level will be measured through the Community Health Activities Model Program for Seniors (CHAMPS) questionnaire.
Depression and anxiety | 8 weeks after surgery
  The Hospital Anxiety and Depression Scale (HADS) will be used to assess anxiety and depression.
Nutritional status | 8 weeks after surgery
  Nutritional status will be assessed using body, body weight loss over the preceding three months (>10%), and/or serum albumin < 35 g -1 will define poor nutritional status. Hand grip strength and body impedance will also be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Carli, MD, Principal Investigator — Montreal General Hospital
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided